CLINICAL TRIAL: NCT00643110
Title: Milk as Treatment for Hypoglycemia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not funded
Sponsor: Creighton University (Other)
Responsible Party: Marc S. Rendell, M.D., Creighton University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rendell 01; Dairy Council - Rendell 01
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Type 1 Diabetes
Keywords: Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: D50 glucose — D50 glucose would be administered, if necessary.

SUMMARY:
Test hypothesis that milk can raise blood sugars as well as orange juice or glucose tablets without raising blood sugars too much the way that orange juice or glucose tablets sometimes do.

DETAILED DESCRIPTION:
Subjects will wear a continuous glucose monitor prior to test to determine normal glucose levels. The morning of the test an IV will be inserted into the subject and insulin and saline drips will be started. Blood glucose levels will be checked every 10 minutes until the subject becomes hypoglycemic. IVs will be stopped at that time and subject will be given skim milk, orange juice or glucose tablets at that time. Blood will be drawn every 15 minutes until blood sugars stabilize. Blood draws will be analyzed to determine glucose, insulin, epinephrine, norepinephrine, glucagon, cortisol, growth hormone and GLP-1 levels. Procedure will be repeated two more times using other glucose methods (skim milk, orange juice or glucose tablets).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes
* Able to be consented
* Able to wear continuous glucose monitor

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Completion of 6 subjects. | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton Diabetes Center, Omaha, Nebraska, United States